CLINICAL TRIAL: NCT01527591
Title: Safety And Long-Term Immunogenicity Of The 13-Valent Pneumococcal Conjugate Vaccine In Children Who Are Solid Organ Transplant Recipients
Brief Title: Pneumococcal Conjugate Vaccine 13 (Prevnar13®) in Children Who Are Solid Organ Transplant Recipients (SOT)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Jaime G. Deville, MD, FAAP, Professor of Clinical Infectious Diseases, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pfizer-Prevnar13®
Record Dates: First submitted 2011-12-21; First posted 2012-02-07 (Estimated); Last update posted 2025-04-02 (Actual); Status verified 2025-01

CONDITIONS: Infection in Solid Organ Transplant Recipients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (1):
- vaccine (Other): pneumococcal conjugated vaccine
  Interventions: Biological: Pneumococcal Conjugate Vaccine 13 (PCV13)

INTERVENTIONS:
Biological: Pneumococcal Conjugate Vaccine 13 (PCV13) — A single intramuscular dose of 0.5 mL.
  Other Names: Prevnar13®

SUMMARY:
The purpose of this study is to determine the safety and long-term immunogenicity of the 13-Valent Pneumococcal Conjugate vaccine in children who are solid organ transplant recipients.

DETAILED DESCRIPTION:
The purpose of this study is to determine if a booster dose of 13-valent pneumococcal conjugate vaccine (PCV13) is safe and results in a measurable and durable immunologic response against pneumococcal subtypes present in the vaccine in solid organ transplant recipient (SOT) children.

Pneumococcal infections are amongst the most common infections seen in immunocompromised children. Infection by Streptococcus pneumoniae is one of the most frequently observed infection in immunocompromised children.

Pneumococcal polysaccharide vaccines (PPV) have been licensed in the U.S. for over 40 years. In contrast, pneumococcal conjugate vaccines are immunogenic and efficacious in normal infants and children, and offer hope of reducing pneumococcal infections in immunocompromised children. However, conjugate pneumococcal vaccine can only protect against a limited number of the 90 pneumococcal serotypes.

It is reasonable to anticipate that the introduction of PCV13 may help reduce the chances of severely immunocompromised children getting pneumococcal infections. Many of these children have been previously immunized with a full series of a 7-valent pneumococcal conjugate vaccine. These children will benefit from an additional dose of the new 13-valent vaccine. The degree to which SOT-recipient children are protected by prior immunizations and are responsive to new immunizations is still largely undefined. This study aims to expand the knowledge regarding the safety and immunogenicity of PCV13 immunization in this growing and vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Are 12 to 59 months of age.
* Have received a solid organ transplantation requiring ongoing immunosuppression.
* Have been receiving immunosuppressive agents for at least 3 months. Non-steroidal anti-inflammatory agents, G-CSF, erythropoietin and inhaled corticosteroids are not considered immunosuppressive agents for the purposes of this study.
* Expect to be able to complete the study injection and follow-up.
* Have parent or guardian's consent.
* Have received at least 3 doses of an approved PCV7 and/or PCV13 vaccine series.

Exclusion Criteria:

* Have received any inactivated vaccine within 4 weeks, or any live vaccine within 6 weeks of entering the study.
* Have had an allergic reaction or a serious side effect after receipt of any previous immunization to pneumococcal vaccines, or to other routine childhood immunizations.
* Have any other condition that would make receiving study vaccine inadvisable.
* Have other diseases of the immune system.
* Have any other disease or previous surgery that would interfere with study treatment.
* Are likely to have bleeding disorders.

Ages: 12 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
To measure antibody concentrations by EIA and opsonophagocytosis assay (OPA) | Measured at different time points until 240 weeks post PCV 13 booster dose
  Immunogenicity, functional antibody responses and sero-conversion will be evaluated by enzyme immunoassay (EIA) and opsonophagocytosis assay to a booster immunization with PCV13 vaccine in SOT-recipient children 12-59 months of age

SECONDARY OUTCOMES:
To measure the extent and persistence of immunity by measuring antibody concentrations by EIA and OPA | Measured at different time points until 240 weeks post PCV 13 booster dose
  To measure the magnitude and persistence of humoral (EIA and OPA) anti--pneumococcal immune responses in children with SOT who were immunized with a booster dose of PCV 13 between 12 and 59 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Jaime G Deville, MD, FAAP, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States